CLINICAL TRIAL: NCT04912778
Title: Profiling of Post Covid-19 Infection Patients: an Online Survey
Acronym: PRESTO
Status: Completed | Type: Observational
Sponsor: Moens Maarten (Other)
Collaborators: STIMULUS research group, Vrije Universiteit Brussel (Unknown)
Responsible Party: Sponsor-Investigator, Moens Maarten, principal investigator, Universitair Ziekenhuis Brussel
Organization: Universitair Ziekenhuis Brussel (Other)
Other Study IDs: PRESTO
Record Dates: First submitted 2021-06-02; First posted 2021-06-03 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Persons who had a covid-19 infection.: Male and female adults who were previously infected with covid-19.
  Interventions: Other: Filling in an online survey

INTERVENTIONS:
Other: Filling in an online survey — Patients are asked to fill in an online survey regarding functional status, quality of life and symptoms of central sensitisation.

SUMMARY:
The aim of this study is to explore the relation between indicators of central sensitisation, quality of life and functional status in patients post covid-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* male and female adults who were previously infected with covid-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study male and female adults who were previously infected with covid-19 will be eligible to complete the survey. No specific criteria will be imposed regarding the time frame after infection.
Sampling Method: Non-Probability Sample
Enrollment: 567 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Functional status | Up to 18 months after infection with Covid-19.
  Post-COVID-19 functional status is evaluated by the Post-COVID-19 Functional Status Scale.
Health-related Quality of life | Up to 18 months after infection with Covid-19.
  The EuroQol with five dimensions and three levels is used to evaluate health-related quality of life.
Symptoms of central sensitisation | Up to 18 months after infection with Covid-19.
  Symptoms of central sensitisation are assessed by the Central Sensitization Inventory.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Belgium

REFERENCES:
- [Derived] Moens M, Duarte RV, De Smedt A, Putman K, Callens J, Billot M, Roulaud M, Rigoard P, Goudman L. Health-related quality of life in persons post-COVID-19 infection in comparison to normative controls and chronic pain patients. Front Public Health. 2022 Oct 20;10:991572. doi: 10.3389/fpubh.2022.991572. eCollection 2022. PMID 36339175